CLINICAL TRIAL: NCT03460925
Title: Interventional Multicentric Study Without Medicine, in Patients Affected by Locally Advanced Pancreatic Adenocarcinoma: Stereotactic Radiotherapy.
Brief Title: Improving REsectability in Pancreatic NEoplasms (IRENE)
Acronym: IRENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRENE-1
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer; Stereotactic Body Radiotherapy
Keywords: pancreatic cancer; stereotactic body radiotherapy; resectability
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT plus chemotherapy (Experimental): Patients with unresectable or "borderline resectable" locally advanced pancreatic carcinoma at time of diagnosis
  Interventions: Radiation: SBRT plus chemotherapy

INTERVENTIONS:
Radiation: SBRT plus chemotherapy — Neoadjuvant stereotactic body radiotherapy (SBRT, 30 Gy in 5 fractions) plus chemotherapy with Folfirinox

SUMMARY:
Evaluation of clinical response in terms of resectability of patients with locally advanced pancreatic cancer treated with neoadjuvant chemotherapy plus stereotactic body radiotherapy.

DETAILED DESCRIPTION:
Aim of the study is to define the percentage of patients with down-staging and clinical response after having undergone stereotactic radiotherapy + chemotherapy with neoadjuvant intent for locally advanced pancreatic carcinoma or "borderline resectable" at the time of diagnosis.

The study evaluates the response to therapy in terms of resectability, of acute and delayed treatment-related toxicity, of overall survival and progression-free survival and also assesses patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of locally advanced pancreatic carcinoma, not upfront surgically treated (according to NCCN resectability criteria), without distant metastases
* NCCN criteria resectability status
* patient's age, performance status, possible presence of comorbidity should also be considered to decide the optimal approach (upfront surgery versus neoadjuvant treatment).
* If the chemotherapy treatment induces the disease to a condition of resectability, the patient will undergo a surgical evaluation
* indication for radiotherapy treatment
* ECOG 0-2
* obtaining informed consent
* not pregnant or breastfeeding

Exclusion Criteria:

* ECOG> 2
* presence of internal diseases for which radiotherapy is contraindicated, or diseases of the connective system, or gastric or duodenal ulcer in progress or acute diverticulitis, ulcerative colitis
* comorbidity which in the opinion of the referring physician may constitute a risk for participation in the study
* lack of availability for clinical-instrumental follow-up
* previous abdominal radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response to the treatment in terms of resectability | 24 months
  Percentage of patients with pancreatic cancer judged to be inoperable who have undergone surgical treatment after neoadjuvant chemotherapy plus stereotactic body radiotherapy. Response is evaluated with CT-scan and 18F FDG PET-scan (RECIST criteria) by a multidisciplinary team of surgeons, radiologist, oncologist, radiation oncologist according to resectability criteria NCCN v. 2017.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Months of survival since the diagnosis
Progression free survival | 24 months
  Progression-free survival (PFS) after radiotherapy is evaluated with CT-scan and 18F FDG PET-scan (RECIST criteria). Also laboratory tests are performed (CA 19.9)
Toxicity | 24 months
  Acute and late toxicities after radiotherapy are assessed with CTCAE v. 4.03
Quality of life | 24 months
  QoL are assessed with Cancer Linear Analog Scale (CLAS) which evaluating well-being, fatigue, and ability to perform daily activities (values range from 0 that represents the best status to 10 that represents the worst one)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Study Director — Radiation Oncology Center, Department of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided